CLINICAL TRIAL: NCT03487679
Title: The Effects of Prolonged Fasting on the Microbiome and HDL Particles of Human Subjects
Brief Title: Effects of Prolonged Fasting on Microbiome and HDL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 918915
Record Dates: First submitted 2018-03-01; First posted 2018-04-04 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Fasting
Keywords: Microbiome; High Density Lipoprotein; Inflammation
MeSH Terms: conditions — Fasting; Inflammation | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fasting (Experimental): Participants will undergo one day of habitual eating followed by 36 hours of water only fasting and final day of habitual eating of the exact same diet consumed on the first eating day. Blood draws will be performed on Day 1 in a 10-12 hr fasted state and 2 hour postprandial state and again on Day 3 in a 36hr fasted state and a 2 hour post prandial state. Microbiome samples and blood glucose data will be collected throughout the course of the study.
  Interventions: Other: Fasting

INTERVENTIONS:
Other: Fasting — Participants will undergo one day of habitual eating followed by 36 hours of water-only fasting and final day of habitual eating consuming the exact same diet consumed on the first eating day. Blood draws will be performed on Day 1 in a 10-12 hr fasted state and 2 hour postprandial state and again on Day 3 in a 36hr fasted state and a 2 hour post prandial state. Microbiome samples and blood glucose data will be collected throughout the course of the study.

SUMMARY:
Participants will undergo one day of habitual eating followed by 36 hours of water only fasting and final day of habitual eating of the exact same diet consumed on the first eating day. Blood draws will be performed on Day 1 in a 10-12 hr fasted state and 2 hour postprandial state and again on Day 3 in a 36hr fasted state and a 2 hour post prandial state. Microbiome samples and blood glucose data will be collected throughout the course of the study.

DETAILED DESCRIPTION:
Screening and Consent:

Prospective subjects who pass the initial phone screening interview (i.e. meet inclusion/exclusion criteria) will be admitted into the study and scheduled for a consent visit. At the consent visit, subjects who decide to participate will be given a series of questionnaires including a health history questionnaire, physical activity questionnaire, and will be asked to complete a 3-day diet record, to be completed before the baseline visit at the beginning of the study. Women who consent to participate will be scheduled to complete the study within the follicular phase and menses of the menstrual cycle to avoid confounding alterations in lipoproteins.

Study Visit1 (Baseline fasted):

On Day 1 of the study protocolstudy participants will report to the Ragle Human Nutrition Research Center located on the UC Davis campus (1283 Academic Surge, University of California, Davis, in Davis CA 95616) for a 12-hour overnight fasting blood draw and anthropometric measurements at approximately 8AM. Any participants that are found to have fasting glucose above or below 70-100mg/dL will be removed from the study. Study participants will be given a Precision Xtra Blood Ketone Testing Kit to collect blood ketone data during the fasting period of the study protocol, a set of stool collection kits to collect stool samples throughout the rest of the study protocoland fitted with a GoBe activity monitor to track physical activity throughout the rest of the study protocol. Proper use, care, and storage of the Precision Xtra systems, stool collection kits, and GoBe monitors will be explained in detail to study participants during the baseline visit. Study participants will be given a 24-hr food diary to record their food and beverage intake throughout the rest of the day or may be asked to track their diet using GB 360.

Study Visit 2 (Baseline postprandial):

After the baseline visit on Day 1 of the study protocol, study participants will go about their normal routines and eat their habitual diet ad libitum while recording their dietary intake throughout the day. This food record will be used in order for the study participants to mimic their food intake on Day 1 during the eating period on Day 3 of the study protocol. Study participants will eat their last meal of the day at approximately 6PM. Post-prandial blood samples will be collected at 2 hours after the ingestion of this last meal and immediately processed to yield patient plasma and isolated PBMCs to be stored for future analysis. These post-prandial samples will constitute the baseline "Fed" state of each participant. Study participants will also perform their first bloodprick for ketone measurement using the Precision Xtra Monitor under instruction and supervision by study personnel.

Fasting:

After ingestion of their final meal, participants will undergo a full 36 hours of fasting comprising Day 2 and the beginning of Day 3 of the trial without otherwise modifying their typical routine, including drinking coffee or tea (but with no creamers or sweeteners of any kind), if this is part of their normal routine. The time of the ingestion of the standardized meal will be used as the start point (0hr) for the continuous 36 hours of fasting. 36 hrs of fasting has been shown to be well tolerated in human subjects and was chosen for this trial as it represents the approximate amount of time that fasting would be experienced during a single cycle of an alternate day fasting regimen. Therefore, results from this study could be generalized to plan for future studies of alternate day fasting. Subjects will be encouraged to report any feelings of dizziness, headaches, nausea, or severe hunger that they may experience and, based on the severity of their conditions, will be advised whether or not to continue with the trial. Subjects will be asked to take small blood pricks starting immediately after waking up on Day 2 and then every 3 conscious hours thereafter using thePrecision Xtra Blood Ketone Testing Kits in order to test blood ketone levels during the fasting period. Ketone levels obtained from the blood pricks will be recorded automatically by the Precision Xtra monitor.

Study Visit 3 (Post 36h fasted):

At 36 hours of fasting, roughly 8AM on Day 3, subjects will return to the Ragle Center, perform a final blood prick for ketone monitoring by the Precision Xtra and their blood samples will be collected and again immediately processed and stored for future analysis constituting the "Fasted" state for each participant.

Study Visit 4 (Post 36h postprandial):

After the blooddraw at Study Visit 3, study participants will be allowed free access to food throughout the rest of the day and asked to eat an identical diet to the dietary intake the participants recorded on Day 1 in their 24 hour food diary. Subjects will eat their last meal at approximately 6PM. Post-prandial blood samples will be collected at 2 hours after the ingestion of this last meal and immediately processed to yield patient plasma and isolated PBMCs to be stored for future analysis. These post-prandial samples will constitute the "Refed" state of each participant. After this final blood draw, the Precision Xtra system will be collected, the GoBe removed, and the activity and ketone data collected throughout the course of the study will be transferred to a secure computer for analysis. Fasting compliance will be determined as 1) increasing or steady ketone levels throughout the 36hr fasting period and 2) the absence of significant drops in blood ketone levels, which would indicate food intake and noncompliance.

StoolCollection (Days 1-3):

Study participants will use the provided stool collection kits to collect stool samples from each bowel movement throughout the entire course of the study. Stool samples will be obtained from study participants at the Ragle Center as soon as possible after initial collection by study participants, frozen, and stored at -80C.

ELIGIBILITY:
Inclusion Criteria:

- Age: 20-40 years old to constitute a young study population; 60-80 years old to constitute an elderly study population

* BMI: 19-27 kg/m2 to constitute a normal/healthy weight population
* Weight: 133lbs or more
* Fasting Glucose: 70-100mg/dL to ensure that fasting can be tolerated without inducing dangerously low levels of blood glucose
* Subjects must be willing to undergo a period of 36 hours of water-only fasting
* Subjects must be willing to collect samples of each bowel movement produced throughout the entire study period for microbiome analysis.
* Subjects must be willing to collect and test blood pricks for blood glucose levels using a Contour Next ONE Blood Glucose Kit during the fasting stage of the study protocol.
* Subjects must be willing to continuously wear a GoBe activity monitor throughout the course of the trial.

Exclusion Criteria:

* Smoker
* Anemia
* Pregnancy or current breast-feeding
* Documented chronic diseases including diabetes, thyroid disease, metabolic syndrome, cancer, or previous cardiovascular events
* Any inflammatory bowel disease including IBS, Crohn's Disease, Celiac Disease
* Consumption of >1 alcoholic drink/day
* Current consumption of any probiotic or prebiotic supplements
* Extreme dietary or exercise patterns
* Recent weight fluctuations (greater than 10% in the last six months)
* Regular use of over-the-counter allergy or pain medications (>1/week)
* Taking prescription lipid medications (e.g. statins) or other supplements known to alter lipoprotein metabolism such as isoflavones.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Change in HDL Immunomodulatory Capacity | Baseline fasted vs. Post 36 hours fasted
  HDL will be isolated from plasma samples and HDL immunomodulatory capacity will be assessed in isolated HDL with an in vitro assay using stimulated macrophages.

SECONDARY OUTCOMES:
Change in Gut Microbiome Composition | Baseline fasted vs. Post 36 hours fasted
  Gut microbial composition will be assessed by sequencing of isolated DNA from stool samples.

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Zivkovic, Ph.D., Principal Investigator — UC Davis
Locations (1):
- University of California Davis, Davis, California, United States

REFERENCES:
- [Derived] Rhodes CH, Zhu C, Agus J, Tang X, Li Q, Engebrecht J, Zivkovic AM. Human fasting modulates macrophage function and upregulates multiple bioactive metabolites that extend lifespan in Caenorhabditis elegans: a pilot clinical study. Am J Clin Nutr. 2023 Feb;117(2):286-297. doi: 10.1016/j.ajcnut.2022.10.015. Epub 2022 Dec 20. PMID 36811567